CLINICAL TRIAL: NCT06673953
Title: Effect of Respiratory Trainer on Cardiopulmonary Functions in Patients with Upper Cross Syndrome Post-Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa ali, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005197
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Post Coronary Artery Bypass Grafting; Post-Cardiac Surgery Patients; Upper Cross Syndrome; Respiratory Muscle Weakness; Respiratory Muscle Training
Keywords: Post-CABG / Upper Cross Syndrome / Respiratory Muscle Training
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Respiratory training (study) group. (Experimental): Thirty patients (n=30) receiving respiratory muscles training and traditional physical therapy program for six weeks (three sessions/ week) for 40-60 minutes.
  Interventions: Other: Respiratory Muscle Training by (The Breather); Other: Traditional physical therapy program
- Traditional (control) group (Active Comparator): Thirty patients (n=30) receiving the traditional physical therapy program for six weeks (three sessions/ week) for 40-60 minutes.
  Interventions: Other: Traditional physical therapy program

INTERVENTIONS:
Other: Respiratory Muscle Training by (The Breather) — Patients are instructed to inhale deeply and forcefully (at non fatigable resistance) for 2-3 seconds, slight pause, and then exhale forcefully for 2-3 seconds for 10 repetitions with 2 sets.
  Other Names: Respiratory Muscle Training
  Arms: Respiratory training (study) group.
Other: Traditional physical therapy program — Traditional physical therapy program in form of: (TENS / Low-intensity continuous ultrasonic / Infrared radiation application / Cervical Stabilization exercise )
  Other Names: Conventional physical therapy program

SUMMARY:
The purpose of this study is to investigate if there is any effect of the respiratory training on cardiopulmonary functions in patients with upper cross syndrome post-cardiac surgery.

Hypothesis:

Null hypothesis: There is no effect of the respiratory training on pulmonary functions in patients with upper cross syndrome post-cardiac surgery.

DETAILED DESCRIPTION:
Sixty post-CABG-male-patients (n=60) with upper cross syndrome, their age ranges from 45 to 55 years old, are selected from Elbank-Elahly hospital (out-patient clinic), Cairo, Egypt. This randomized control study is performed after assessing and randomly assigning patients, (through using a computer program which generates random numbers), into two equal groups (30 patients for each group).

Respiratory training (study) group. Thirty patients (n=30) will receive respiratory muscles training and traditional physical therapy program for six weeks (three sessions/ week) for 40-60 minutes.

Traditional (control) group. Thirty patients (n=30) will receive the traditional physical therapy program for six weeks (three sessions/ week) for 40-60 minutes.

All subjects enrolled in the study are informed about the aim, technique, and experimental protocol of this study before participation. A written informed consent is assigned before participation.

After open-heart surgeries, patients with median sternotomy must restrict upper limbs movements that stretch the sternum, for 8 to 12 weeks after surgery, and avoid raising their arms above the head.

In addition, inappropriate posture such as forward head posture caused by the incision leads to upper cross syndrome. This causes an inability to perform activities of daily living, and chronic neck pain which adversely affects the respiratory system due to respiratory muscle imbalance.

Chronic neck pain (CNP), due to upper cross syndrome, is one of the most prevalent and costly musculoskeletal complaints associated with significant functional disability.

Equipment:

A. Evaluative equipment:

1. Weight and height scales: To measure body weight and height to calculate BMI.
2. Visual Analog Scale (VAS): To assess pain severity.
3. Pressure biofeedback instrument: To measure endurance of deep cervical flexors (DCF).
4. Electronic Spirometer: Digital-CONTEC-SP10-Spirometer-Lung-Breathing-Diagnostic-Vitalograph-Spirometry-Model CMS501 (Made in China), to measure ventilatory function test parameters.

   Forced expiratory volume in the first second (FEV1), Forced vital capacity (FVC), FEV1/FVC ratio. and Peak expiratory flow rate (PEFR).
5. Pittsburgh Sleep Quality Index. To measure sleep quality (Arabic version)
6. pulse oximetry. To measure HR, and SPO2 (Pulse Oximeter GRANZIA Model No: AS-304).
7. Sphygmomanometer: To measure ABP (Model Number: GT001-110/111 aneroid sphygmomanometer, Zhejiang, China)
8. Stopwatch. To measure six-minute walk test time.
9. Short Form 36 (SF-36) Health Survey Questionnaire: To measure quality of life.

B. Treatment equipment:

1. Respiratory muscle trainer device (The Breather device).
2. DCF muscles training device: Pressure biofeedback (Stabilizer TM, Chattanooga Group, Inc., Chattanooga, TN)
3. Gymna electrotherapy device.
4. EME ultrasound-therapy device.
5. A 650-W infrared halogen lamp (Philips Electronics Industries)

Procedure:

A. Evaluation Procedures: All patients will follow the same evaluative procedures before (baseline) and after 12 weeks of treatment. (illustrated in the Outcome Measures section)

B. Therapeutic procedures:

Respiratory training (study) group: Patients will receive:

1. Respiratory muscles training: They will be asked to perform respiratory training through The Breather device beginning with the easiest setting. They will be instructed to inhale deeply and forcefully (at non fatigable resistance) for 2-3 seconds, slight pause, and then exhale forcefully for 2-3 seconds for 10 repetitions with 2 sets.
2. Traditional physical therapy program in the form of:

   * TENS: Conventional TENS will be applied at high frequency (from 50 Hz to 130 Hz), low intensity (comfortable, not painful) and small pulse duration (50 μs to 200 μs). By applying small surface electrodes on the neck paraspinal muscles for 20 minutes.
   * Low-intensity continuous ultrasonic waves will be applied on the neck paraspinal muscles (trigger points of the trapezius muscles) for 10 minutes.
   * Infrared radiation application will be used for 10 minutes: The lamp should cover the area over the upper back and neck regions.
   * Cervical Stabilization exercise will be performed after three repetitions of stretching exercises for neck muscles as warm-up and cool-down exercises. Then, the exercise will be executed in supine position; the cuff will be put suboccipital. They will reach a 5mm Hg pressure target with increments of 2 mm Hg from a baseline of 20mm Hg to the ultimate level of 30mm Hg with hold for 10 seconds. The duration of contraction will gradually increase up to 10 seconds for each target level. Subjects will perform ten repetitions before progressing to the next target level.

Traditional (control) group: Patients will receive the traditional physical therapy program.

ELIGIBILITY:
Inclusion Criteria:

* Sixty post-CABG-male-patients for at least three months and their age ranges from 45 to 55 years old.
* Craniovertebral angle < 51°, but not less than 30°.
* Non-specific chronic neck pain: defined as neck pain without an identifiable pathological cause and attributed to poor posture without radiation to upper limbs.
* VAS score between 3-7.
* Their body mass index ranges from (25 -29.9) kg/m2.
* Values of FEV1 and FVC lower than 80%

Exclusion Criteria:

* Rheumatoid arthritis, cervical disc pathology, and traumatic neck pain.
* History of respiratory disease and clinical signs of severe cardiac events.
* Neurological disorders which affect the diaphragm.
* Patients whose BMI is less than 25, or greater than 30 kg/m2.
* Smokers.
* Values of FEV1 and FVC higher than 80%
* Patients with chronic obstructive pulmonary disease or asthma.

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 60 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Pulmonary functions: | Baseline (assessment), and at 12 weeks post-intervention.
  Measurements of ventilatory function are recorded before and after receiving the treatment sessions (FEV1, FVC, FEV1/FVC, MVV).
  Assessing respiratory improvement.
  Unit of Measure: Liters (L)
Six-Minute-Walk Test | Baseline (assessment), and at 12 weeks post-intervention.
  Patients are asked to walk for 6 minutes along a flat corridor. Measured in meters, assessing exercise capacity and functional improvement.
  The SpO2 and heart rate are measured continuously during testing.
  Heart Rate (HR): Measured in beats per minute (BPM), evaluating cardiovascular response.
  SpO2 (Peripheral Oxygen Saturation): Assessing: Blood oxygen saturation levels to evaluate respiratory and cardiovascular efficiency. Unit of Measure: Percentage (%)
VO2 max (Maximal Oxygen Consumption) | Baseline (assessment), and at 12 weeks post-intervention.
  Assessing: Maximum oxygen uptake during high-intensity exercise to evaluate aerobic capacity and cardiopulmonary function.
  Estimated based on an equation which contains:
  weight is body weight (kg), 6MWD is distance walked in 6 min (m), age (years), BMI is calculated body mass index(kg/m2), height is body height (cm) and HR is heart rate at the end of the walking test.
  Unit of Measure: mL/kg/min
Pittsburgh Sleep Quality Index. | Baseline (assessment), and at 12 weeks post-intervention.
  Respondents are asked to indicate how frequently they have experienced certain sleep difficulties and rate them. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Short Form 36 (SF-36) Health Survey Questionnaire (Arabic version). | Baseline (assessment), and at 12 weeks post-intervention.
  A 36-item scale measures eight domains of health status. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Pain severity | Baseline (assessment), and at 12 weeks post-intervention.
  Assessing intensity of perceived pain for monitoring changes in pain severity throughout the intervention. Pain severity is assessed by the self-reported Visual Analog Scale (VAS). By using a 10 cm line where patients mark their pain level, with 0 representing "no pain" and 10 representing "worst imaginable pain." Unit of Measure: Points on a 0-10 scale
Endurance of DCF | Baseline (assessment), and at 12 weeks post-intervention.
  Endurance of DCF muscles is measured by a pressure biofeedback instrument. The patient lays in the crook lying position and the pressure biofeedback instrument is placed under the neutral cervical spine below the occiput and inflated up to 20 mmHg. The subjects perform this movement at 5 different pressure levels, i.e., 22, 24, 26, 28, and 30 mmHg. Each level is supposed to be held for 10 sec, and the test terminated if they are unable to hold the position for 10 sec at any level or if the maximum level is achieved (30 mmHg).
Craniovertebral angle measurement | Baseline (assessment), and at 12 weeks post-intervention.
  Adhesive markers are placed on the tragus of the right ear and the C7 spinous process, and the subjects are instructed to stand by side (lateral view) and to look at a target in front of them with both arms beside the body. Then, a digital camera is fixed at the level of the 7th cervical vertebra. Finally, the Surgi map Spine software is used to analyze the digitalized photographs and measure CVA. It is the angle between 2 imaginary lines: the horizontal line passing through the spinous process of C7 and the line passing from C7 to the tragus of the ear.
Weight and height measurement | Baseline (assessment)
  Weight and height are recorded, and BMI will be calculated according to the formula: BMI = Weight (Kg) / Height (m2)

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Helmy, Professor, Study Chair — Professor of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics. Faculty of Physical Therapy. Cairo University; El-Sayed Felaya, Lecturer, Study Director — Lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics. Faculty of Physical Therapy. Cairo University; Ahmed Elsisi, Assistant Professor, Study Director — Assistant Professor of Critical Care Medicine. Faculty of Medicine. Beni suef University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Giza Governorate, Egypt